CLINICAL TRIAL: NCT01555983
Title: The Effect of Vaporized Cannabis on Neuropathic Pain in Spinal Cord Injury
Brief Title: Vaporized Cannabis and Spinal Cord Injury Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Barth Wilsey (Other)
Collaborators: VA Northern California Health Care System (U.S. Federal Agency); University of California, San Diego (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Barth Wilsey, Research Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 256412; 1R01DA030424-01A1 (NIH)
Record Dates: First submitted 2012-02-09; First posted 2012-03-16 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-02

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: cannabis; central neuropathic pain; analgesia
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Marijuana Abuse; Agnosia | interventions — Medical Marijuana

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vaporization of Cannabis 6.7% THC (Active Comparator): Inhaling of standardized measured puffs of Vaporized High Dose 6.7% THC. Monitored for 8 hours measuring psychoactive and analgesic effects.
  Interventions: Drug: Vaporization of Cannabis
- Vaporization of Cannabis 2.9% THC (Active Comparator): Inhaling standardized measured puffs of Vaporized Low Dose 2.9% THC. Monitored for 8 hours measuring psychoactive and analgesic effects.
  Interventions: Drug: Vaporization of Cannabis
- Vaporization of Cannabis Placebo THC (Placebo Comparator): Inhaling standardized measured puffs of Placebo THC. Monitored for 8 hours measuring psychoactive and analgesic effects.
  Interventions: Drug: Vaporization of Cannabis

INTERVENTIONS:
Drug: Vaporization of Cannabis — Randomized, Controlled Crossover Trial of Vaporized Cannabis using different strengths of THC in patients with Central Neuropathic Pain Active Comparator: Vaporized High Dose 6.7% THC Active Comparator: Vaporized High Dose 2.9% THC Placebo Comparator: Vaporized Placebo THC
  Other Names: Medical Marijuana

SUMMARY:
This study will demonstrate that vaporized marijuana results in antinociception when compared to placebo in subjects with spinal cord injury. To further evaluate potential benefits and side effects, the effect of different strengths of cannabis on mood, cognition, and psychomotor performance will also be measured.

DETAILED DESCRIPTION:
This study will demonstrate that vaporized cannabis can produce antinociceptive effects compared to placebo in human subjects with spinal cord injury (SCI). A within-subject crossover study of the effects of cannabis versus placebo on spontaneous and evoked pain will be performed. A synopsis of antinociception with mood, cognitive impairment, psychomotor performance, and side effects will be obtained to help evaluate the utility of vaporized marijuana in SCI neuropathic pain.

This study will compare the analgesic and side effect profile of low (3.5%) to high dose (7.0%) delta 9-tetrahydrocannabinol in subjects with spinal cord injury pain. It is hypothesized that a low dose will produce a lesser degree of neuropsychological impairment while maintaining a similar degree of pain relief to the higher dose. The use of two different strengths will help determine tolerable dosing for the treatment of SCI neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 and less than 70
2. Pain intensity ≥ 4/10
3. Neuropathic pain defined as chronic pain in an area of sensory abnormality corresponding to the spinal cord or nerve root lesion, and the pain should have no primary relation to movement, inflammation or other local tissue damage
4. Leeds Assessment of Neuropathic Symptoms and Signs score greater than or equal to 12
5. Spinal cord injury of 3 or more months duration (to avoid spontaneous recovery obfuscating generalizability)

Exclusion Criteria:

1. Known concomitant cerebral damage/cognitive impairment (TBI, Alzheimer's Disease Vascular dementia, Parkinson's disease, dementia with Lewy Bodies and Front temporal dementia
2. Clinically significant or unstable medical condition (i.e., cardiac, respiratory, hepatic or renal disease) that, in the opinion of the investigator, would compromise participation in the study
3. Neurologic disorders unrelated to spinal cord injury that may confound the assessment of the central neuropathic pain due to spinal cord injury (hereditary neuropathies; diabetic peripheral neuropathy; traumatic neuropathy; and immune-mediated neuropathies)
4. Active substance abuse within past year using "The Substance Abuse Module of Diagnostic Interview Schedule for DSM-IV
5. Pregnancy as ascertained by a self-report and a mandatory commercial pregnancy test
6. Currently on probation or parole.
7. Hx of Schizophrenia, Bipolar Depression with Mania, current suicidal ideation or past history of suicide attempt 8. Severe depression (Patient Health Questionnaire-9 ≥ 15) 9. Current suicidal ideation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barth Wilsey, MD, Principal Investigator — UC San Diego, Department of Psychiatry
Locations (1):
- UC Davis CTSC Clinical Research Center , Sacramento VA Medical Center, Mather, California, United States

IPD SHARING:
Plan to Share IPD: Yes
email Barth Wilsey at bwilsey@ucsd.edu

REFERENCES:
- [Background] Wilsey B, Marcotte T, Tsodikov A, Millman J, Bentley H, Gouaux B, Fishman S. A randomized, placebo-controlled, crossover trial of cannabis cigarettes in neuropathic pain. J Pain. 2008 Jun;9(6):506-21. doi: 10.1016/j.jpain.2007.12.010. Epub 2008 Apr 10. PMID 18403272
- [Background] Abrams DI, Jay CA, Shade SB, Vizoso H, Reda H, Press S, Kelly ME, Rowbotham MC, Petersen KL. Cannabis in painful HIV-associated sensory neuropathy: a randomized placebo-controlled trial. Neurology. 2007 Feb 13;68(7):515-21. doi: 10.1212/01.wnl.0000253187.66183.9c. PMID 17296917
- [Background] Abrams DI, Vizoso HP, Shade SB, Jay C, Kelly ME, Benowitz NL. Vaporization as a smokeless cannabis delivery system: a pilot study. Clin Pharmacol Ther. 2007 Nov;82(5):572-8. doi: 10.1038/sj.clpt.6100200. Epub 2007 Apr 11. PMID 17429350
- [Background] Ellis RJ, Toperoff W, Vaida F, van den Brande G, Gonzales J, Gouaux B, Bentley H, Atkinson JH. Smoked medicinal cannabis for neuropathic pain in HIV: a randomized, crossover clinical trial. Neuropsychopharmacology. 2009 Feb;34(3):672-80. doi: 10.1038/npp.2008.120. Epub 2008 Aug 6. PMID 18688212
- [Background] Wallace M, Schulteis G, Atkinson JH, Wolfson T, Lazzaretto D, Bentley H, Gouaux B, Abramson I. Dose-dependent effects of smoked cannabis on capsaicin-induced pain and hyperalgesia in healthy volunteers. Anesthesiology. 2007 Nov;107(5):785-96. doi: 10.1097/01.anes.0000286986.92475.b7. PMID 18073554

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled via recruitment from the UC Davis Medical Center Spinal Cord Injury Clinic, IRB-approved recruitment letters and newspaper advertisements.
Pre-assignment Details: Screening for inclusion criteria (e.g., age > 18 and ≤ 70, pain intensity ≥ 4/10 and Leeds Assessment of Neuropathic Symptoms and Signs, a pain scale based on analysis of sensory description and bedside examination of sensory dysfunction. A threshold of ≥12 on this instrument was utilized to substantiate neuropathic pain.
Groups:
- Placebo First, Then 2.9%THC, Then 6.7% THC: Placebo in am of first intervention visit, 2.9%THC in am of second intervention visit (after 3-10 day washout period) and then 6.7%THC in am of third intervention visit (after 3-10 day washout period).
- Placebo First, Then 6.7%THC, Then 2.9%THC: Placebo in am of first intervention visit, 6.7%THC in am of second intervention visit (after 3-10 day washout period) and then 2.9%THC in am of third intervention visit (after 3-10 day washout period).
- 2.9%THC First, Then Placebo, Then 6.7%THC: 2.9%THC in am of first intervention visit, placebo in am of second intervention visit (after 3-10 day washout period) and then 6.7%THC am of third intervention visit (after 3-10 day washout period)
- 2.9%THC First, Then 6.7%THC, Then Placebo: 2.9%THC in am of first intervention visit, then 6.7%THC in am of second intervention visit (after 3-10 day washout period) and then placebo in am of third intervention visit (after 3-10 day washout period).
- 6.7%THC First, Then Placebo, Then 2.9%THC: 6.7%THC in am of first intervention visit, then placebo in am of second intervention visit (after 3-10 day washout period) and then 2.9%THC in am of third intervention visit (after 3-10 day washout period).
- 6.7%THC First, Then 2.9%THC, Then Placebo: 6.7%THC in am of first intervention visit, then 2.9%THC in am of second intervention visit (after 3-10 day washout period) and then placebo in am of third intervention visit (after 3-10 day washout period).
Period: Overall Study
Arm/Group | Placebo First, Then 2.9%THC, Then 6.7% THC | Placebo First, Then 6.7%THC, Then 2.9%THC | 2.9%THC First, Then Placebo, Then 6.7%THC | 2.9%THC First, Then 6.7%THC, Then Placebo | 6.7%THC First, Then Placebo, Then 2.9%THC | 6.7%THC First, Then 2.9%THC, Then Placebo
Started | 9 | 7 | 7 | 7 | 5 | 7
Completed | 8 (One subject only finished the placebo session, then dropped out of study) | 7 | 7 | 7 | 4 (One subject complete 6.7%THC and placebo sessions, then dropped out) | 6 (One subject completed the 6.7%THC session, then dropped out.)
Not Completed | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Consented subjects with at least one study visit
Groups:
- All Study Participants: All participants received all interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Reduction in Pain Intensity of 30% or More
Description: Number of participants achieving a reduction of pain intensity of 30% or more, a level believed to be clinically important, was estimated for each treatment dose.
Time Frame: hourly pain assessments for 8 hours
Measure: Number; unit: participants
Groups:
- Placebo THC: Session at which placebo THC was administered
- 2.9% THC: Vaporization of Cannabis 2.9% THC
- 6.7% THC: Vaporization of Cannabis 6.7% THC
Arm/Group | Placebo THC | 2.9% THC | 6.7% THC
Number analyzed (Participants) | 41 | 38 | 41
participants | 18 | 26 | 35
Statistical Analysis 1: Comparison: Placebo THC vs 2.9% THC vs 6.7% THC; The number needed to treat (NNT) to achieve 30% pain reduction during the 8-hour period was 4 (95% CI: 2.1-25.3) for the lower dose vs. placebo, and 3 (95% CI: 1.6-4.2) for the higher dose versus placebo; Test type: Superiority or Other; p < .05, Mixed Models Analysis; Cochran-Armitage trend tes = .0001

ADVERSE EVENTS:
Time Frame: participants were followed for the 8 hour duration of clinical research center stay
Groups:
- Placebo THC: Vaporization of Cannabis Placebo THC
Arm/Group | Placebo THC | 2.9% THC | 6.7% THC
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38 | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo THC (N=41) | 2.9% THC (N=38) | 6.7% THC (N=41)
orthostatic hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Patient had orthostatic hypotension. Symptomatically, he stated he was going to "pass out" and the the room went dark. BP initially unobtainable but returned to baseline with assuming supine position.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No